CLINICAL TRIAL: NCT05286866
Title: Comparison Between High-speed Drilling With Irrigation and Low-speed Drilling: a Randomized Clinical Trial
Brief Title: Comparison Between High-speed Drilling With Irrigation and Low-speed Drilling With Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Juan Carlos Bernabeu Mira (Unknown); Miguel Peñarrocha Diago (Unknown)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Titular Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1937615
Record Dates: First submitted 2022-02-17; First posted 2022-03-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Bone Loss
Keywords: dental implant; low speed; irrigation; drilling
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low speed drilling without irrigation (Experimental): The dental implants will be placed using a low-speed drilling technique without irrigation for the experimental group.
  Interventions: Procedure: Dental implant bed preparation
- High speed drilling with irrigation (Active Comparator): The dental implants will be placed using a high-speed drilling technique with irrigation for the control group.
  Interventions: Procedure: Dental implant bed preparation

INTERVENTIONS:
Procedure: Dental implant bed preparation — Drilling an osteotomy for placement of a dental implant

SUMMARY:
A randomized controlled clinical trial was conducted in the Oral Surgery Unit, Faculty of Medicine and Dentistry, University of Valencia. The research was carried out following the principles described in the Helsinki Declaration and the study was approved by the Institutional Review Board of the Ethics Committee of the University of Valencia (1937615).

Fifty patients were included in the study according to the selection criteria.The osteotomies were randomized in two groups: the control group was performed under the high-speed drilling (800 rpm) with irrigation technique and the study group under the low-speed drilling without irrigation technique (50 rpm). The randomization tool was www.randomization.com.

DETAILED DESCRIPTION:
Before the intervention, a preoperative orthopantomography and CBCT (Cone Beam Computerized Tomography) were taken for all the patients. Every patient was submitted a prophylactic hygiene 7 days before the intervention and 2 g of oral amoxicillin tablet 1 hour before the intervention (Clamoxyl®, GlaxoSmithKline, Madrid, Spain) was prescribed as a prophylaxis medication.

All the surgeries were performed by the same experienced operator (JCBM). The interventions were conducted under local anesthesia (4% articaine with 1: 100,000 adrenaline (Inibsa®, Lliça de Vall, Barcelona, Spain). The IPX® implant model (Nueva Galimplant S.L, Sarria, Galicia, Spain) was placed in the present study.

Surgical drills with stop (K Fres Stop ®, Nueva Galimplant S.L, Sarria, Spain) were used to prepare the osteotomies. The drilling sequence used will be: initial lance drill, followed by conical drills of 2.0 mm, 2.6 mm, 3.2 mm and 3.6 mm. The implants were apico-coronally situated at 4 mm to the mucosal margin with a torque of 35 Ncm.

The placed implants were IPX Model (Nueva Galimplant S.L., Sarria, Spain) with a 2-mm height anti-rotational abutment of one piece (Nueva Galimplant S.L, Sarria, Spain). The healing was non-submerged.

As postoperative medication 1 g of paracetamol (Bexistar®, Bacino Laboratory, Barcelona, Spain) on demand maximum every 8 hours were prescribed. Postoperative hygiene and oral care instructions were explained to the patient. A mouthwash of 0.12% chlorhexidine (GUM®, John O. Butler / Sunstar, Chicago, IL, USA) twice daily for two weeks was recommended too. The sutures were removed 7 days after surgery. Prosthetic loading will be performed 10 weeks after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults, plaque and bleeding index less than 25%, sufficient bone height and width for implant placement, vestibular keratinized gingiva of at least 2 mm and stable occlusion and healthy periodontium.

Exclusion Criteria:

* any edentulous area requiring bone grafting procedures, medical conditions that contraindicate implant surgery such as severe bruxism or poor hygiene, pregnant or lactating patients, bisphosphonate therapy, patients receiving chemotherapy and radiotherapy to the head and neck, patients non-collaborators, incomplete data collection or lack of control assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Evaluation the marginal bone loss around the dental implants | 12 months follow-up
  Measurement of peri-implant bone loss in millimeters through a periapical radiograph

SECONDARY OUTCOMES:
Calculation of the elapsed drilling time | 1 day
  Drilling time calculation in seconds
Analysis of the bone harvesting | 1 day
  Calculation of the harvested bone between the flutes of the surgical drills in grams
Evaluation of the patient satisfaction (pressure, distress, time, vibration and anguish) | 1 day
  Measurement of the pressure, distress, time, and vibration using a visual analog scale (VAS). The minimum value is "0" (nothing) and maximum value is "100" (the most one imaginable).
Evaluation of the quality of life (mouth opening, chewing, speaking, sleeping, daily routine and work) | 7 days
  Measurement of the mouth opening, chewing, speaking, sleeping, daily routine and work through a Likert Scale. 0= nothing, 1=little bit, 2=something/sometimes, 3=Quite, 4=a lot.
Analysis of the postoperative pain through a visual analog scale (VAS) | 7 days
  Measurement of postoperative pain through a visual analog scale (VAS). The minimum value is "0" (no pain) and maximum value is "100" (the worst pain imaginable)
Evaluation of the peri-implant soft tissue | 12 months follow-up
  Probing depth measurement in millimeter (mm) using a periodontal probe
Analysis of the postoperative inflammation | 7 days
  Measurement of postoperative inflammation through a visual analog scale (VAS). The minimum value is "0" (no inflammation) and maximum value is "100" (the worst inflammation imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Odontología de la Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernabeu-Mira JC, Penarrocha-Diago M, Canullo L, Camacho-Alonso F, Rojo-Sanchis J, Penarrocha-Oltra D. Peri-Implant Marginal Bone Changes Using High-Speed Drilling With Irrigation Versus Low-Speed Drilling Without Irrigation: A Randomized Clinical Trial With 12 Months of Follow-Up. Clin Oral Implants Res. 2025 Jun;36(6):698-709. doi: 10.1111/clr.14416. Epub 2025 Feb 14. PMID 39950686